CLINICAL TRIAL: NCT05599386
Title: Predictors of Acute and Persistent Postoperative Pain in Lung Cancer Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jannie Bisgaard Stæhr (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor-Investigator, Jannie Bisgaard Stæhr, Chief Physician, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: AAUH-VATS-02
Record Dates: First submitted 2022-10-24; First posted 2022-10-31 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Undergoing VATS: Only one group as primary endpoints are continous
  Interventions: Diagnostic Test: Preoperative test

INTERVENTIONS:
Diagnostic Test: Preoperative test — Patients are subject to quantitative sensory testing, questionnaires, and biomarker analysis prior to surgery.

SUMMARY:
The aim of this observational study is to investigate if preoperative quantitative sensory testing, anxiety and depression symptoms, and biological markers are associated with the risk of developing acute and chronic postoperative pain after video-assisted Thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
This observational study examine acute and chronic postoperative pain in patients undergoing VATS. In the study preoperative biomarkers, quantitative sensory testing and questionnaires are used to create prediction models for acute and chronic postoperative pain. The study will serve as background information on the risk factors and predictive factors as well as an exploration of the impact of surgical stress from VATS on circulation microRNA and inflammatory mediators.

ELIGIBILITY:
Inclusion Criteria:

* Adults independent of sex with an age of ≥ 18 years
* Patients scheduled for VATS as a part of either examination or radical treatment of lung cancer

Exclusion Criteria:

* Patients who are unable to understand oral and written information.
* Patients with known chronic pain in the thorax which have been persisting for at least six months before the day of surgery.
* Pregnant and nursing women.
* Patients receiving a planned preoperative epidural blockade during their stay.
* Patients converted to open surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Public University hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2024-08-06 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | 48 hours postoperative
  Pain intensity on a Numerical Rating Scale ranging from 0 indicating no pain to 10 indicating worst pain imaginable during the first two postoperative days.
Numerical Rating Scale | 365 days postoperative
  Pain intensity on a Numerical Rating Scale ranging from 0 indicating no pain to 10 indicating worst pain imaginable at follow up. Collected using the Brief Pain Index

SECONDARY OUTCOMES:
Total equipotent opioid dose | Total equipotent opioid dose in milligrams during the first 48 hours after surgery.
  48 hours postoperative
Time to first administration of opioid | Time in hours to first postoperative administration of Pro Re Nata (PRN) opioids
  48 hours postoperative
Mobilisation | 48 hours postoperative
  Time in hours to full mobilisation defined as walking with or without aids.
Patient-reported satisfaction of postoperative pain management assessed by self-made questionnaire in Danish | Measured twice. Once 48 hours after surgery or at non fixed time(on average 4 days and a maximum of 3 months) as well as at 365 days
  Patients are asked to fill out a questionnaire rating their general satisfaction with pain management and sufficiency of pain treatment on a scale from 0 to 10. The questionnaire also assess whether the patients had any perceived side effects and how uncomfortable they were on a scale from 0 to 10.

OTHER OUTCOMES:
Examination of the level of inflammatory biomarkers (IL-6, IL-8, TNFa, etc.) and circulation microRNA | 48 hours postoperative
  Change in expression of microRNA and Inflammatory mediators from before surgery until two days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jannie Bisagaard, MD, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Region of Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No